CLINICAL TRIAL: NCT00804089
Title: Randomised Comparative Pragmatic Clinical Trial of Traditional Acupuncture and Superficial Dry Needling and Acupressure of Myofascial Trigger Points for the Treatment of Patients With Chronic Mechanical Low Back Pain
Brief Title: Traditional Acupuncture and Myofascial Trigger Point Dry Needling and Acupressure for Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hermano Miguel Foundation (Other)
Collaborators: Ecuadorian Federation of Physiotherapy, Tungurahua Branch (Unknown); Technical University of Ambato (Other)
Responsible Party: Sergiy Voznesenskyy, Ph.D., B.P.T., Hermano Miguel Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AR1-001-2008
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Low Back Pain
Keywords: Low Back Pain, Chronic; Acupuncture; Dry Needling; Acupressure; Acupuncture Points; Trigger Points, Myofascial
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Traditional needle acupuncture
  Interventions: Procedure: Traditional needle acupuncture
- 2 (Active Comparator): Myofascial trigger point dry needling
  Interventions: Procedure: Myofascial trigger point dry needling
- 3 (Active Comparator): Myofascial trigger point acupressure
  Interventions: Procedure: Myofascial trigger point acupressure

INTERVENTIONS:
Procedure: Traditional needle acupuncture — Traditional needle acupuncture using traditional meridian acupoints and Ashi (tender) points
  Arms: 1
Procedure: Myofascial trigger point dry needling — Superficial dry needling of myofascial trigger points found in the muscles related to low back pain, followed by their postisometric stretching
  Arms: 2
Procedure: Myofascial trigger point acupressure — Blunt needle acupressure of myofascial trigger points found in the muscles related to low back pain, followed by their postisometric stretching
  Arms: 3

SUMMARY:
The purpose of this study is to compare the therapeutic effects of acupuncture using traditional acupoints and Ashi points with myofascial trigger points superficial dry needling and acupressure, followed by postisometric stretching of the appropriate muscles, in the treatment of patients with chronic mechanical low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mechanical lower back pain for at least three months.
* The chronic mechanical lower back pain is the chief complaint, with or without leg pain.
* The lower back pain is disabling to the degree that affects the patient's routine job and/or his or her lifestyle.

Exclusion Criteria:

* Patients with tumor, infection, major trauma to the spine causing fracture or disruption of the major ligaments, or cauda equina syndrome.
* Patients with neurological signs of spinal nerve compression.
* Patients having undergone spinal surgery, facet joint block and/or corticoid injection.
* Patients with general contraindications for acupuncture or acupressure treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sergiy Voznesenskyy, Ph.D. B.P.T., Principal Investigator — Hermano Miguel Foundation
Locations (2):
- Ecuador (2):
  - Social Security Hospital, Ibarra, Imbabura
  - Social Security Hospital, Ambato, Tungurahua Province